CLINICAL TRIAL: NCT01362621
Title: A 2-year Prospective, Multi-center, Observational and Epidemiologic Outcomes Study of the Disease Course and Unmet Needs in Children With Symptomatic Moderate to Severe Allergic Asthma
Brief Title: Observational and Epidemiologic Study of the Disease Course and Unmet Needs in Children With Symptomatic Moderate to Severe Allergic Asthma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Other Study IDs: CIGE025BUS26
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Moderate to Severe Allergic Asthma
Keywords: Allergic asthma; Pediatrics; Exacerbations; Perennial aeroallergens; Inhaled corticosteroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood sample was collected at either screening (Visit 1) or enrollment (Visit 2). These samples were collected for DNA extraction. The extracted DNA is stored at Novartis Pharmaceuticals Corporation for pharmacogenetic analysis and storage.

GROUPS / COHORTS (1):
- Children 6 to less than 12 years of age

SUMMARY:
The study was designed to collect data about inadequately controlled moderate to severe allergic asthma in subjects 6 to < 12 years of age, managed in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Total IgE ≥30 IU (historical values obtained within 3 months of screening visit will be accepted). If historic result not available, to be obtained at screening visit.
* Diagnosis of asthma for at least 12 months prior to screening visit date, or symptoms compatible with asthma for at least 12 months if diagnosis made within 12 months of screening visit
* Documented sensitivity to one or more perennial aeroallergens as evidenced by a positive skin prick test or in-vitro specific IgE test for dust mites, cat dander, dog dander or cockroach within the preceding one year of the screening visit
* Prescribed inhaled corticosteroid for at least 3 months prior to screening (A) and having evidence of inadequately controlled disease either with at least one from list (B) OR history of asthma-related exacerbations as defined in (C). [e.g., A and (B or C)]

A. Fluticasone DPI > 200 mcg/day or equivalent ex-valve dose ICS, or if ≤ 200 mcg fluticasone DPI or equivalent plus another daily controller medication (i.e. LABA, leukotriene antagonist or theophylline)

B. At least one of the following in the preceding 4 weeks prior to the screening visit:

* on average asthma symptoms > 2 days/week or multiple times in a day on ≤ 2 days/week
* nighttime awakenings ≥ 2 times/month due to asthma symptoms
* use of SABAs > 2 times/week on average
* some limitation in activity due to asthma
* on spirometric evaluation, FEV1 ≤ 80% of predicted, FEV1/FVC ≤ 80%, or peak expiratory flow rate ≤ 80% of personal best

C. Minimum of 2 asthma exacerbations requiring oral corticosteroid bursts in the 12 months previous to the screening visit

Exclusion Criteria:

* Subjects currently enrolled in a clinical study of a therapeutic agent or biologic agent or who participated in a clinical study of a therapeutic agent within 30 days of Visit 1 or a biologic agent within 120 days of Visit 1
* Subjects with a history of prior use of omalizumab
* Subjects with a severe medical condition that in the view of the investigator prohibits participation in the study by either impairment in the ability to answer questions or follow instructions (e.g., severe neurological or developmental disorder)
* Subjects with serious respiratory-related medical conditions other than allergic asthma such as, but not limited to, allergic bronchopulmonary aspergillosis, cystic fibrosis or bronchiectasis
* Subjects with elevated serum IgE levels for reasons other than allergy such as, but not limited to, parasitic infections, hyperimmunoglobulin E syndrome, and Wiskott-Aldrich Syndrome

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6 to less than 12 years old with moderate to severe allergic asthma for at least 12 months, treated with inhaled corticosteroids for at least 3 months but remaining symptomatic
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The change from basline in Childhood Asthma Control Test | 2 years
The change from baseline in total Wasserfallen Clinical Symptom Score | 2 years

SECONDARY OUTCOMES:
The change from baseline for overall score in the Standardized Pediatric Asthma Quality of Life Questionnaire (PAQLQ(S)) | 2 years
The change from baseline for overall score in Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) | 2 years
The number of days of missed school. | 2 years
The number of days of missed work. | 2 years

CONTACTS AND LOCATIONS:
Locations (51):
- United States (50):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Crescent City, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Roseville, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Thornton, Colorado
  - Novartis Investigative Site, Albany, Georgia
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Columbus, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Cynthiana, Kentucky
  - Novartis Investigative Site, Metarie, Louisiana
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Stevensville, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Plymouth, Minnesota
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Berkeley Heights, New Jersey
  - Novartis Investigative Site, Brick, New Jersey
  - Novartis Investigative Site, Summit, New Jersey
  - Novartis Investigative Site, West Orange, New Jersey
  - Novartis Investigative Site, Batavia, New York
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Rockville Centre, New York
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Gresham, Oregon
  - Novartis Investigative Site, Allentown, Pennsylvania
  - Novartis Investigative Site, Altoona, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, South Burlington, Vermont
  - Novartis Investigative Site, Emporia, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Bellingham, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, San Juan, Puerto Rico